CLINICAL TRIAL: NCT01969825
Title: The Role of Massage in Increasing Total Motile Sperm Count of Intrauterine Insemination
Brief Title: The Role of Massage in Increasing Total Motile Sperm Count of IUI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Massage2013
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2013-10

CONDITIONS: Infertility
Keywords: Infertility; Intrauterine insemination; Male factor infertility; Massage; Total motile sperm count
MeSH Terms: conditions — Infertility | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Massage (Experimental): Professional Swedish massage less than 15 minutes prior to semen collection for intrauterine insemination.
  Interventions: Behavioral: Massage
- No massage (No Intervention): Normal protocol for semen collection prior to intrauterine insemination.

INTERVENTIONS:
Behavioral: Massage
  Arms: Massage

SUMMARY:
The purpose of this prospective, randomized study, was to determine if neck and shoulder massage performed within 15 minutes of semen sample collection will increase the semen volume, and therefore increase the total motile sperm available for insemination as a result of decreased stress.

ELIGIBILITY:
Inclusion Criteria:

* Infertility,
* initiating clomiphene + IUI therapy
* signed study consent

Exclusion Criteria:

* Severe male infertility (baseline semen concentration < 10 million total motile sperm)
* female bilateral tubal occlusion
* failure to ovulate with clomiphene
* failed clomiphene + IUI therapy (three prior cycles with no conception)
* unable to tolerate clomiphene
* unable or unwilling to follow study protocol

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Total Motile Sperm Count | 1 month
  The primary outcome variable is total motile sperm count, which is determined based on the semen volume, concentration, and motility.

SECONDARY OUTCOMES:
Pregnancy | 3 months
  Pregnancy rate per cycle with intrauterine insemination.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Hurst, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Women's Institute at Carolinas Medical Center, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Gerhard I, Lenhard K, Eggert-Kruse W, Runnebaum B. Clinical data which influence semen parameters in infertile men. Hum Reprod. 1992 Jul;7(6):830-7. doi: 10.1093/oxfordjournals.humrep.a137745. PMID 1323572
- [Background] Cui KH. The effect of stress on semen reduction in the marmoset monkey (Callithrix jacchus). Hum Reprod. 1996 Mar;11(3):568-73. doi: 10.1093/humrep/11.3.568. PMID 8671268
- [Background] Jurewicz J, Hanke W, Sobala W, Merecz D, Radwan M. [The effect of stress on the semen quality]. Med Pr. 2010;61(6):607-13. Polish. PMID 21452563
- [Background] Giblin PT, Poland ML, Moghissi KS, Ager JW, Olson JM. Effects of stress and characteristic adaptability on semen quality in healthy men. Fertil Steril. 1988 Jan;49(1):127-32. doi: 10.1016/s0015-0282(16)59663-0. PMID 3335259
- [Background] Fenster L, Katz DF, Wyrobek AJ, Pieper C, Rempel DM, Oman D, Swan SH. Effects of psychological stress on human semen quality. J Androl. 1997 Mar-Apr;18(2):194-202. PMID 9154514
- [Background] Collodel G, Moretti E, Fontani V, Rinaldi S, Aravagli L, Sarago G, Capitani S, Anichini C. Effect of emotional stress on sperm quality. Indian J Med Res. 2008 Sep;128(3):254-61. PMID 19052335
- [Background] De Souza MJ, Arce JC, Pescatello LS, Scherzer HS, Luciano AA. Gonadal hormones and semen quality in male runners. A volume threshold effect of endurance training. Int J Sports Med. 1994 Oct;15(7):383-91. doi: 10.1055/s-2007-1021075. PMID 8002116
- [Background] McGrady AV. Effects of psychological stress on male reproduction: a review. Arch Androl. 1984;13(1):1-7. doi: 10.3109/01485018408987495. PMID 6152527
- [Background] Sefton JM, Yarar C, Berry JW. Six weeks of massage therapy produces changes in balance, neurological and cardiovascular measures in older persons. Int J Ther Massage Bodywork. 2012;5(3):28-40. doi: 10.3822/ijtmb.v5i3.181. Epub 2012 Sep 26. PMID 23087776
- [Background] Moyer CA, Rounds J, Hannum JW. A meta-analysis of massage therapy research. Psychol Bull. 2004 Jan;130(1):3-18. doi: 10.1037/0033-2909.130.1.3. PMID 14717648
- [Background] Hodgson NA, Lafferty D. Reflexology versus Swedish Massage to Reduce Physiologic Stress and Pain and Improve Mood in Nursing Home Residents with Cancer: A Pilot Trial. Evid Based Complement Alternat Med. 2012;2012:456897. doi: 10.1155/2012/456897. Epub 2012 Jul 24. PMID 22888364
- [Background] Reindollar RH, Regan MM, Neumann PJ, Levine BS, Thornton KL, Alper MM, Goldman MB. A randomized clinical trial to evaluate optimal treatment for unexplained infertility: the fast track and standard treatment (FASTT) trial. Fertil Steril. 2010 Aug;94(3):888-99. doi: 10.1016/j.fertnstert.2009.04.022. Epub 2009 Jun 16. PMID 19531445
- [Background] Moyer CA, Seefeldt L, Mann ES, Jackley LM. Does massage therapy reduce cortisol? A comprehensive quantitative review. J Bodyw Mov Ther. 2011 Jan;15(1):3-14. doi: 10.1016/j.jbmt.2010.06.001. Epub 2010 Jul 2. PMID 21147413
- [Background] Thirthalli J, Naveen GH, Rao MG, Varambally S, Christopher R, Gangadhar BN. Cortisol and antidepressant effects of yoga. Indian J Psychiatry. 2013 Jul;55(Suppl 3):S405-8. doi: 10.4103/0019-5545.116315. PMID 24049209
- [Background] Huang W, Taylor A, Howie J, Robinson N. Is the diurnal profile of salivary cortisol concentration a useful marker for measuring reported stress in acupuncture research? A randomized controlled pilot study. J Altern Complement Med. 2012 Mar;18(3):242-50. doi: 10.1089/acm.2010.0325. Epub 2012 Mar 2. PMID 22385023